CLINICAL TRIAL: NCT02233660
Title: Changes in Function, Cervical Range of Motion and Pinch Grip Force After Physical Therapy in Carpal Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: The Role of the Cervical Spine in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUFA PI -12/0023
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Carpal Tunnel Syndromes
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy Group. (Experimental): The physical therapy group will receive 3 treatment sessions of manual therapies including maneuvers targeted to the areas anatomically related to the median nerve (i.e., cervical spine, shoulder, elbow and wrist) of 30min of duration, once per week.
  Interventions: Other: Physical Therapy Group
- Surgical Group (Active Comparator): The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Interventions: Procedure: Surgical Group

INTERVENTIONS:
Other: Physical Therapy Group — The physical therapy group will receive 3 treatment sessions of manual therapies including maneuvers targeted to the areas anatomically related to the median nerve (i.e., cervical spine, shoulder, elbow and wrist) of 30min of duration, once per week.
  Arms: Physical Therapy Group.
Procedure: Surgical Group — The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Arms: Surgical Group

SUMMARY:
This randomized clinical trial will investigate changes in hand function, active cervical range of motion and pinch grip force after the application of physical therapy in women with carpal tunnel syndrome (CTS). The purpose of this study is to compare changes in function, cervical range of motion and pinch grip force induced after the application of a physical therapy program including manual therapies targeted to those areas related to the median nerve or after endoscopic surgery in women with CTS at medium and long-term follow-up. The hypothesis is that manual therapy is more effective for increasing cervical range of motion and pinch grip force, but similarly effective for improving function, than surgical treatment in women with CTS.

DETAILED DESCRIPTION:
There is some evidence suggesting that CTS is associated with restricted cervical range of motion and deficits in pinch grip force. In fact, restricted cervical range of motion and deficits in pinch grip force seems to be independent of electro-diagnostic findings. These findings would be associated with the proposed "double crush syndrome" theory. However no longitudinal studies have been conducted. Further it has been demonstrated that hand function is associated to deficits in these outcomes. Since previous studies support the use of physical therapy and surgical interventions for the management of function in these patients, the aim of this study is to conduct a randomized clinical trial to determine if changes in hand function are related to changes in active cervical range of motion and pinch grip force after the application of a physical therapy program including manual therapies targeted to those areas related to the median nerve or endoscopic surgery in women with CTS.

ELIGIBILITY:
Inclusion Criteria:

* Pain and paresthesia in the median nerve distribution
* Positive Tinel sign,
* Positive Phalen sign,
* Symptoms had to have persisted for at least 6 months
* Deficits of sensory and motor median nerve conduction according to guidelines of the American Association of Electrodiagnosis, American Academy of Neurology, and the American Physical Medicine and Rehabilitation Academy

Exclusion Criteria:

* Any sensory/motor deficit related to the ulnar or radial nerve;
* Older than 65 years of age;
* Previous surgical intervention, steroid injections or physical therapy intervention
* Multiple diagnoses of the upper extremity (eg, cervical radiculopathy);
* History of neck, shoulder, or upper limb trauma (whiplash);
* History of any systemic disease causing CTS (eg, diabetes mellitus or thyroid disease);
* History of other systemic conditions (eg, rheumatoid arthritis, fibromyalgia);
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in hand function between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used to assess function. This questionnaire evaluates 2 domains: 1) the functional status scale assesses ability to perform 8 common hand-related tasks; and, 2) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5-point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity. In the current study the score of the functional status scale of this questionnaire will be used as the main outcome.

SECONDARY OUTCOMES:
Changes in active cervical range of motion between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention
  A cervical range of motion (CROM) device will be used to assess cervical range of motion in a single direction: flexion, extension, lateral flexion toward or away from the side of the CTS, and rotation toward or away from the side of the CTS. For patients with unilateral symptoms, sides are classified as affected or unaffected whereas in those with bilateral symptoms, the most painful side will be considered as the affected side and the less painful side as the unaffected side.
Changes in pinch grip force between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention
  Pinch grip force between the tip of the thumb with the tip of the index or the little finger will be measured with a pinch grip dynamometer

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Fundación Alcorcon, Alcorcón, Madrid
  - Universidad Rey Juan Carlos, Alcorcón, Madrid

REFERENCES:
- [Derived] Fernandez-de-Las-Penas C, Cleland J, Palacios-Cena M, Fuensalida-Novo S, Pareja JA, Alonso-Blanco C. The Effectiveness of Manual Therapy Versus Surgery on Self-reported Function, Cervical Range of Motion, and Pinch Grip Force in Carpal Tunnel Syndrome: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Mar;47(3):151-161. doi: 10.2519/jospt.2017.7090. Epub 2017 Feb 3. PMID 28158963